CLINICAL TRIAL: NCT06316544
Title: China Elderly Comorbidity Medical Database
Acronym: CECMed
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Hongwei Li, MD, Professor, Beijing Friendship Hospital
Other Study IDs: CECMed; 2021ZD0111000 (Other Grant/Funding Number: National Science and Technology Major Project)
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease; Hypertension; Diabetes Mellitus; Osteoporosis; COPD Chronic Obstructive Pulmonary Disease
Keywords: elderly; Comorbidity; Chronic diseases
MeSH Terms: conditions — Coronary Artery Disease; Hypertension; Diabetes Mellitus; Osteoporosis; Pulmonary Disease, Chronic Obstructive; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this observational cohort study is to provide comprehensive evaluation and early warning for elderly patients with chronic diseases. The main question it aims to answer is: How to explore effective evaluation methods for diseases in elderly patients based on the coexistence of multiple diseases and high individual heterogeneity? How to explore the key indicators and influencing factors of adverse events in elderly patients.. Participants will be followed up at 1, 3, 6, 9, and 12 months to obtain adverse event information.

DETAILED DESCRIPTION:
Older people represent the fastest growing sector of society and account for the largest increase in hospital admissions. They are at highest risk of acquired disability, cognitive decline, or admission to residential care, either as a consequence of illness or as an unfortunate consequence of treatment. Older people's needs are more complex with potentially coexistent medical, functional, psychological, and social needs.At the same time, comorbidities among the elderly are also extremely common, which resulting in clinical medical decision-making complex and difficult. The comorbidity rate among elderly people in the community is 76.5%; The comorbidity rate of elderly hospitalized patients can reach 91.3%. Hypertension, diabetes, coronary heart disease, COPD and osteoporosis are five common chronic diseases. Because of the intersection of risk factors, the occurrence of comorbidity is particularly obvious. In addition, frailty, malnutrition and other geriatric syndromes also seriously affect the prognosis of elderly patients with chronic diseases. The treatment plans for elderly comorbidities are often contradictory and conflicting. Medical decision-making is complex and difficult. Traditional specialized disease diagnosis and treatment benefits are limited, and the risk of iatrogenic problems is high, which further consuming medical resources. Therefore, in order to further improve the prognosis of elderly patients with chronic diseases, we established a cohort for the above five chronic disease patients, searched for risk factors for adverse events, explored effective methods for evaluating elderly patients with chronic diseases, and improved their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years old;
* At least one of hypertension, type 2 diabetes, coronary heart disease, osteoporosis, chronic obstructive pulmonary disease (COPD). Coronary heart disease: Heart disease caused by stenosis or occlusion of the official cavity caused by coronary atherosclerosis, resulting in myocardial ischemia, hypoxia or necrosis. This includes chronic myocardial ischemic syndrome (stable angina, ischemic cardiomyopathy, and occult coronary heart disease) and acute coronary syndrome (unstable angina and acute myocardial infarction). type 2 diabetes: HbA1c is greater than 6.5% or fasting blood glucose is greater than 126mg/dL (7.0mmol/L), and fasting is defined as no calorie intake for at least 8 hours; Or oral glucose tolerance test (OGTT) with blood glucose levels greater than 200mg/dL (11.1mmol/L) within 2 hours; Or clinical manifestations of hyperglycemia, random blood glucose greater than 200mg/dL (11.1mmol/L); Or is/has been using hypoglycemic drugs/insulin therapy. Hypertension: Twice random blood pressure, systolic blood pressure (SBP) higher than 140mmHg and/or diastolic blood pressure (DBP) higher than 90mmHg; Or is/has been taking antihypertensive medication. Chronic obstructive pulmonary disease: There are COPD related risk factors and respiratory symptoms, and lung function suggests that there is still airflow restriction after inhaling bronchodilators. The first second forced expiratory volume/forced vital capacity (FEV1/FVC) is less than 0.7. Osteoporosis: A metabolic bone disease characterized by decreased bone mass, destruction of bone tissue microstructure, increased bone fragility, and susceptibility to fractures. The diagnostic criteria are as follows: 1. A history of brittle fractures; 2. When there is no fracture, relying on dual energy X-ray absorption examination method: when measuring the axial bone density or the bone density T value of the hip or distal 1/3 of the radius is less than -2.5, it can be considered as osteoporosis.

Exclusion Criteria:

* Late stage malignant tumors, expected survival time less than 3 months;
* Completely disabled and unable to communicate;
* Unable to cooperate with follow-up.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The included patients are elderly (aged ≥ 65 years) patients with chronic diseases, including coronary heart disease, hypertension, diabetes, COPD, osteoporosis. One of the five common chronic diseases of the elderly, and patients who meet the diagnosis of one of the above five diseases will be include.
Sampling Method: Probability Sample
Enrollment: 4100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Pneumonia/pulmonary infection | 1, 3, 6, 9, 12 months
respiratory failure | 1, 3, 6, 9, 12 months
pulmonary encephalopathy | 1, 3, 6, 9, 12 months
acute exacerbation of chronic obstructive pulmonary disease | 1, 3, 6, 9, 12 months
unstable angina pectoris | 1, 3, 6, 9, 12 months
acute myocardial infarction | 1, 3, 6, 9, 12 months
acute hemorrhagic stroke | 1, 3, 6, 9, 12 months
acute ischemic stroke | 1, 3, 6, 9, 12 months
acute heart failure/acute exacerbation of chronic heart failure | 1, 3, 6, 9, 12 months
malignant ventricular arrhythmia | 1, 3, 6, 9, 12 months
sudden death | 1, 3, 6, 9, 12 months
falls | 1, 3, 6, 9, 12 months
fractures | 1, 3, 6, 9, 12 months
gastrointestinal bleeding | 1, 3, 6, 9, 12 months
pulmonary embolism | 1, 3, 6, 9, 12 months
deep vein thrombosis | 1, 3, 6, 9, 12 months
diabetes ketoacidosis | 1, 3, 6, 9, 12 months
diabetes hyperosmolar coma | 1, 3, 6, 9, 12 months
rehospitalization | 1, 3, 6, 9, 12 months
  any cause of rehospitalization
admission to ICU | 1, 3, 6, 9, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China